CLINICAL TRIAL: NCT05935397
Title: HanYang University Medical Center (HYUMC) PCI Registry
Brief Title: HanYang University Medical Center (HYUMC) Registry
Acronym: HYUMC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Hanyang University (Other)
Responsible Party: Principal Investigator, Young-Hyo Lim, Prof., Hanyang University Seoul Hospital
Other Study IDs: HYUMC
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Stenosis; Coronary Artery Disease; Blood Pressure
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- patients with CAD undergoing PCI: patients with CAD undergoing PCI with second generation DES
  Interventions: Device: percutaneous coronary intervention

INTERVENTIONS:
Device: percutaneous coronary intervention — patients with CAD undergoing PCI with second generation DES

SUMMARY:
The HYUMC registry is a two-center, real-world registry of percutaneous coronary intervention in patients with coronary artery disease. From January 2012, PCI-treated patients from Hanyang University Seoul Hospitals and Hanyang University Guri Hospitals were enrolled in this registry.

The aim of this registry is to examine the long-term clinical outcomes and identify predictors of adverse outcomes following percutaneous coronary intervention conducted at academic hospitals.

DETAILED DESCRIPTION:
In the HYUMC registry, the researchers have gathered and assessed various demographic, laboratory, echocardiographic, and angiographic measurements (both on-admission and during follow-up), as well as conducted questionnaires among patients who underwent percutaneous coronary intervention. The primary focus of this registry is to examine the effects of these parameters on long-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients with CAD who underwent PCI one or more drug eluting stent (DES) with from 2012 at the Division of Cardiology of Hanyang University Seoul Hospital and Hanyang University Guri Hospital, Korea.

Exclusion Criteria:

* second or subsequent hospitalization records of patients with multiple admissions
* patients who died during index hospitalization
* patients who treated with first-generation drug eluting stent
* patients with an outpatient follow-up record of less than 6 months
* patients with insufficient medical records.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with CAD
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MACCE (major adverse cardiac and cerebrovascular event) | 10-year
  the composite of all-cause death, myocardial infarction, stroke, or any revascularization

SECONDARY OUTCOMES:
All-cause death | 10-year
  death from any cause
Myocardial infarction, | 10-year
  presence of clinical symptoms with the presence of electrocardiographic changes, or imaging evidence of new loss of viable myocardium or new regional wall motion abnormalities, in conjunction with elevated levels of cardiac biomarker above the 99th percentile upper reference limit
Stroke | 10-year
  neurological deficit resulting from acute focal damage to the central nervous system due to a vascular cause, requiring hospitalization, and confirmed by a neurologist through imaging findings
Any revascularization | 10-year
  PCI or coronary artery bypass surgery on either target or nontarget vessels

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Hanyang University Guri Hospital, Guri-si
  - Hanyang University Seoul Hospital, Seoul
  - Young-Hyo Lim, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Kim BS, Lim YH, Shin J, Shin JH. Association of systolic blood pressure target and variability with long-term clinical outcomes in patients undergoing percutaneous coronary intervention. Clin Hypertens. 2025 Apr 1;31:e13. doi: 10.5646/ch.2025.31.e13. eCollection 2025. PMID 40201318
- [Derived] Kim BS, Shin JH, Kim W, Kook H, Lee Y, Park JK, Shin J, Lim YH. Association of office blood pressure with ischemic and bleeding events in patients undergoing percutaneous coronary intervention. Sci Rep. 2024 Sep 2;14(1):20310. doi: 10.1038/s41598-024-71060-8. PMID 39218965